CLINICAL TRIAL: NCT04811937
Title: Development of a Computer-aided Polypectomy Decision Support
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was abandoned due to the Covid pandemic which prevented recruitment.
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20.382
Record Dates: First submitted 2021-02-16; First posted 2021-03-23 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Adenomatous Polyps
Keywords: Polyps detection; Artificial Intelligence; Adenoma detection; Polyps classification; Computer decision support
MeSH Terms: conditions — Adenomatous Polyps

STUDY DESIGN:
Intervention Model Description: prospective, multi-endoscopist, single center, clinical study at tertiary referral center (CHUM)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Artificial intelligence for real-time Computer decision support of resection of colorectal polyps (Experimental): A standard colonoscopy will be performed according to the standard of routine care. All optically diagnosed polyps will be removed and sent to the CHUM pathology laboratory for histopathological evaluation according to institutional standards. The AI system will capture video of the procedure in real time, and provide additional information about polypectomy procedures.
  Interventions: Diagnostic Test: Computer-aided polypectomy decision support by Artificial Intelligence

INTERVENTIONS:
Diagnostic Test: Computer-aided polypectomy decision support by Artificial Intelligence — The AI system will capture the live video of the procedure and the AI feedbackwill be shown on a second screen installed next to the regular endoscopy screen. Screen A will show the regular endoscopy image and screen B will show the regular endoscopy image together with the areas that might harbor a polyp and the information to help the polypectomy.

SUMMARY:
Quality components of colonoscopy include the detection and complete removal of colorectal polyps, which are precursors to CRC. However, endoscopic ablation may be incomplete, posing a risk for the development of "interval cancers". The investigators propose to develop a solution based on artificial intelligence (AI) (CADp computer-aided decision support polypectomy) to solve this problem.This research project aims to develop CADp, a computer decision support solution (CDS) for the ablation of colorectal polyps from 1 to 20 mm.

DETAILED DESCRIPTION:
This research project aims to develop CADp, a computer-based decision support (CDS) solution for the removal of colorectal polyps ranging from 1-20 mm. The investigators will use a video and image dataset of polypectomy procedures to train the CADp model; thus, it can provide real-time overlaid video feedback for polypectomy procedures based on five specific metrics: 1) estimation of polyp size; 2) prediction of morphology and histology; 3) suggestion of an appropriate resection accessory and technical approach based on the characteristics, size, and histology of the polyp according to current guidelines; 4) image overlay, based on semantic image segmentation technology, showing the extent of the lesion and suggestion of an appropriate resection margin contour around the polyp to ensure its complete removal; 5) post-resection analysis to identify any remnant polyp tissue or insufficient resection margin that may increase this risk.

The investigators will collect a set of images and video data from live polypectomy procedures to leverage recent advances in AI technology to train deep learning models. This dataset will be obtained prospectively from a cohort of adults (ages 45-80) undergoing screening, diagnostic, or surveillance colonoscopies. To train the CADp solution, the investigators will obtain the corresponding completeness of resection status using the yield of post-resection margin biopsies. The dataset will be divided into two groups, the training, and the CADp test, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age 45-80 years
* Indication to undergo a lower GI endoscopy.

Exclusion Criteria:

* Known inflammatory bowel disease
* Active colitis
* Coagulopathy
* Familial polyposis syndrome;
* Poor general health, defined as an American Society of Anesthesiologists (ASA) physical status class >3
* Emergency colonoscopies

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the CADp system | 3 weeks
  accuracy with which the CADp system predicts completeness of polypectomy in the test set with the reference standard for completeness being determined by the histology of post-polypectomy margin biopsies; if free from any polyp tissue (adenomatous, serrated or hyperplastic), the resection will be considered complete. If remnant polyp tissue is detected in any one or more of the margin biopsies the resection is deemed incomplete
Completeness of polypectomy | 1 month
  We will evaluate the agreement between the different subjective and objective ways of assessing the completeness of the polypectomy : evaluation of margins (presence or not, measurement of margins) by endoscopists self-assessment, and by expert consensus.
Training CADp | 1 month
  Evaluation of the concordance of data on polyp size, extension of margins around the polyp, quality of resection between clinical data (endoscopists' self-assessment and experts' assessments) and CADp prediction.
Validity of the choice of primary outcome | 1 month
  Based on the results and comparison of the different assessment methods, we will perform sensitivity analyses to assess the validity and robustness of the choice of primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel von Renteln, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier Universitaire de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No